CLINICAL TRIAL: NCT04641078
Title: Stereotactic Body Radiotherapy With or Without Darolutamide for OligoRecurrent Prostate Cancer: a Randomized Phase II Trial (DART)
Brief Title: Stereotactic Body Radiotherapy With or Without Darolutamide for OligoRecurrent Prostate Cancer
Acronym: DART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-06863
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer; Prostate Cancer Recurrent; Prostate Cancer Metastatic; Metastatic Cancer; Oligometastasis
Keywords: Radiotherapy; Metastasis-directed therapy; Oligometastatic recurrent hormone sensitive prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): SBRT + 6 months of darolutamide (600 mg b.i.d.)
  Interventions: Drug: Darolutamide; Radiation: metastasis-directed treatment
- Arm B (Other): SBRT only
  Interventions: Radiation: metastasis-directed treatment

INTERVENTIONS:
Drug: Darolutamide — 600 mg BID
  Arms: Arm A
Radiation: metastasis-directed treatment — stereotactic body radiotherapy

SUMMARY:
The current trial will test the combination of darolutamide with SBRT, in oligometastatic recurrent hormone sensitive prostate cancer. We hypothesize that the addition of short-term darolutamide improves metastasis-free survival when added to SBRT without a detrimental impact on the QoL. Considering the large reluctance of both patients and physicians to be randomized to observation, we propose to use the historical data from previous reported randomized trials (STOMP and ORIOLE) as a comparator to explore as a secondary endpoint.

DETAILED DESCRIPTION:
As of the 2018 EAU guidelines, PSMA PET-CT is now recommended for prostate cancer patients with a rising PSA following local therapy, resulting in an increase in patients with conventional imaging M0, but novel imaging M1-state. This creates a new class of patients for which no clear guidelines exist on the optimal management. It became clear that there is no real consensus nor data on how these patients should be treated.

In 1995, a new approach was proposed, hypothesizing that patients with a limited number of metastases (oligometastases) might benefit from eradication of metastases by means of local therapy, or metastasis-directed therapy. Stereotactic body radiotherapy (SBRT), a novel radiotherapy technique for metastatic and primary prostate cancer treatments, has emerged as a highly precise radiotherapy method able to eradicate small metastases with acceptable toxicity. Nevertheless, responses following SBRT were not always durable. To improve response rates and time to new metastases, additional steps should be taken balancing with potential added toxicity. One of the logical steps would be to combine SBRT with temporary androgen deprivation therapy (ADT) as this combination therapy is standard of care for primary PCa and locally recurrent PCa17. However, ADT, negatively impacts quality of life (QoL) even when used temporary. Anti-androgen or androgen receptor (AR) pathway inhibitors (ARpI) may circumvent these side effects by suppressing AR transcription by competitive inhibition of AR, without lowering systemic testosterone. The current trial will test the combination of darolutamide with SBRT, in oligometastatic recurrent hormone sensitive prostate cancer. We hypothesize that the addition of short-term darolutamide improves metastasis-free survival when added to SBRT without a detrimental impact on the QoL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven initial diagnosis of adenocarcinoma of the prostate
* Biochemical relapse of PCa following radical local prostate treatment (radical prostatectomy (RP), primary radiotherapy or the combination of RP and prostate bed adjuvant/ salvage radiotherapy) according to the EAU guidelines 2018.
* Following RP, patients with a biochemical relapse are eligible in case a metastatic relapse is detected even in the absence of prior postoperative prostate bed radiotherapy (adjuvant or salvage). In the absence of prior prostate bed radiotherapy, prostate bed radiotherapy is mandatory for all pT3a or higher or patients with a positive margin at time of RP.
* For patients without prior RP that have a suspected local recurrence following primary radiotherapy, a biopsy should confirm local recurrence. Patients with a confirmed local recurrence and metastases are eligible in case they also undergo a local salvage therapy.
* Metastatic relapse on PSMA PET-CT with a maximum of 5 metastases (any M1a, M1b or M1c). Concomitant diagnosis of N1 disease is allowed as long as all lesions are treated with SBRT and the total number of lesions does not exceed 5. PSMA positive lesions will be scored using the MI-RADS scoring system with lesions scored 4 or 5 considered positive19.
* Asymptomatic for metastatic PCa
* Age >= 18 years
* WHO class 0-1
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given in accordance with to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Local relapse in the prostate gland or prostate bed not suitable for a local salvage treatment
* Small cell carcinoma of the prostate
* PSA doubling time >12 months
* Serum testosterone level <50ng/dl or 1.7 nmol/L at time of randomization
* Currently receiving ADT or PSA rise while on active treatment with ADT (LHRH-agonist, LHRH-antagonist, anti-androgen or estrogen) within the past 6 weeks
* Spinal cord compression or impending spinal cord compression
* Metastases in previously irradiated areas precluding safe delivery of SBRT
* Contraindications to darolutamide
* Previous treatment with cytotoxic agent for PCa
* Treatment during the past month with products known to influence PSA levels (e.g. fluconazole, finasteride, corticosteroids,…)
* Other active malignancy, except non-melanoma skin cancer or other malignancies with a documented disease-free survival for a minimum of 3 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | 2 year
  Metastasis-free survival is defined as time between randomization and the appearance of a new metastatic recurrence (any M1) as suggested by PET-CT or death due to any cause.

SECONDARY OUTCOMES:
Clinical progression-free survival | 2 year
  Clinical progression-free survival is defined as the time between randomization and the appearance of a new lesion (any N1 or M1), a local recurrence as suggested by PET-CT, symptoms related to progressive PCa, or death due to any cause.
Biochemical relapse-free survival | 2 year
  For patients who had previous RP at initial diagnosis, a biochemical recurrence is defined by any confirmed PSA rise above 0.20 ng/ml with a confirmatory rise at least 2 weeks later. For patients who had previous RT to the prostate at initial diagnosis, a biochemical recurrence is defined as the nadir + 2ng/ml (Phoenix definition). Non-responders are considered to have a biochemical recurrence in case a second measurement at least 2 weeks later confirms a rising PSA
Time to next systemic therapy | 4 year
  Time to next systemic therapy is defined as the initiation of any PCa systemic treatment. Systemic therapy will typically be initiated on progression and/or development of new metastases, but indications are at the discretion of the physician.
Castrate resistant-free survival | 4 year
  Time to castration resistant disease is defined as the time from trial randomization until castration resistant status
Prostate cancer-specific survival | 4 year
  PCa-specific survival will be read as the time from trial randomization to the date of death due to PCa.
Overall survival | 4 year
  Overall survival will be read as the time from trial randomization to the date of death from any cause.
Toxicity: acute toxicity | 3 months
  Radiotherapy toxicity will be assessed according to NCI CTCAE v5.0.
Toxicity: late toxicity | 2 year
  Radiotherapy toxicity will be assessed according to NCI CTCAE v5.0.
Patient reported QOL as per EORTC-QLQ C30 | 2 year
  Validated questionnaire assessing different health-related parameters (psychological, physical and social well-being) in cancer patients. A higher score of a symptom scale or item indicates a worse condition; a higher score of a functional scale or global health status/QoL indicates a better condition. A clinically meaningful change is defined as a change from baseline of at least 10 points (i.e., about one-half standard deviation) in either direction.
Patient reported QOL as per EORTC-QLQ PR25 | 2 year
  Validated questionnaire assessing the health-related QOL of prostate cancer patients. A higher score of a symptom scale or item indicates a worse condition; a higher score of a functional scale or global health status/QoL indicates a better condition. A clinically meaningful change is defined as a change from baseline of at least 10 points (i.e., about one-half standard deviation) in either direction.

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (8):
- Belgium (8):
  - OLVZ Aalst, Aalst
  - GZA, Antwerp
  - AZ St-Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - AZ St-Lucas Gent, Ghent
  - Ghent University Hospital, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk